CLINICAL TRIAL: NCT03895710
Title: Longitudinal Associations Between Changes in Sleep Duration and Blood Pressure Across School Holiday in Sleep-deprived Teenagers
Brief Title: Changes in Sleep Duration and Blood Pressure Across School Holiday in Teenagers
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Albert Martin Li, Prof, Chinese University of Hong Kong
Other Study IDs: CREC2015.701
Record Dates: First submitted 2019-03-26; First posted 2019-03-29 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Sleep Deprivation
Keywords: sleep duration; blood pressure; adolescents; holiday
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva samples will be collected with Salivette tubes for assessing the level of cortisol and cortisone, as a reflection of stress which on its own can influence both sleep pattern and BP.
  Participants will be asked to collect their saliva in the morning when they are wearing the BP monitor. Each subject will have to provide five saliva samples according to a fixed sampling protocol: (1) one hour before bedtime, (2) immediately after awakening, (3) 15 min after awakening, (4) 30 min after awakening, and (5) 45 min after awakening.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sleep-deprived group: i. Self-reported time in bed (period from bedtime to get-up time) during school days of <8 hours per day ii. Self-perceived insufficient sleep during school days
- Normal sleep group: i. Self-reported time in bed during school days of >=8 hours per day ii. Self-perceived sufficient sleep during school days

SUMMARY:
Our research question is: Are changes in sleep duration that occur naturally over school holidays associated with changes in blood pressure (BP) in sleep-deprived adolescents?

In this study, the investigators will take advantage of changes in sleep duration that occur during school holidays in adolescents who are sleep deprived (>6 months' history of sleeping <8 hours per night during school term). The investigators will monitor the changes in ambulatory BP and sleep duration over a period of 3 weeks which consist of a week at school, followed by a week of holiday when natural sleep extension takes place, and then another week of school after the holiday. Sleep-wake cycle will be recorded throughout the whole study period with actigraphy and sleep diary. Twenty-four hour ambulatory BP monitoring will be performed on the same weekday during each study week, when salivary cortisol will also be collected. The primary outcome measure is the difference in ambulatory BP parameters between school term and holiday. A control group without sleep deprivation (history of sleeping >8 hours per night) will also be studied concurrently

It is hypothesized that changes in sleep duration are negatively associated with changes in BP. If this study confirms our hypothesis, sleep extension can be used as a relatively inexpensive and simple behavioural intervention in the management and prevention of blood pressure abnormalities. More importantly positive results from this project will provide background information on which government and local school policy can be based and altered for the betterment of our youths.

DETAILED DESCRIPTION:
This is a cohort study that consists of 4 visits over a 3-week study period that includes two periods of 7-day school attendance and one period of 7-day school holiday (Study design flow chart). Subjects who have undergone physical examination and completed the screening questionnaire, and are found to meet all the inclusion and none of the exclusion criteria will be recruited. The first study week will be during school days, followed by a week of school holiday, and the final week is when the subject returns back to school after the holiday. The 3 periods need not to be consecutive so as to allow more flexibility to cater for the subjects' schedule. All assessments however have to be completed within 60 days to minimize the effects of growth on BP / sleep pattern.

Screening

During screening examination, participants will undergo a series of anthropometric measurements. The body build of the subject will be assessed using standard procedures. Standing height (in metres) will be measured without shoes using a Harpenden Stadiometer (Holtain, UK). Body weight will be measured by an electronic weighing scale (Tanita BF-522, Japan). Waist and hip circumference (in centimetres) will also be obtained. Body mass index and waist circumference will be converted into z score using local reference. Blood pressure will be taken using the Datascope Accutorr Plus. Two measurements are taken at 1-minute intervals, with a third reading taken 5 minutes later if the difference between the first two >4 mmHg. The average of two repeatable readings (difference ≤4 mmHg) will be used. Sexual maturity rating will be evaluated by a validated gender specific self-assessment questionnaire. Subjects will have to fill in a sleep questionnaire asking about their sleep habits and symptoms, pediatric daytime sleepiness scale (PDSS), Epworth sleepiness scale (ESS), and strength and difficulties questionnaire (SDQ). Information on parental medical history will also be obtained from the parents using a medical history questionnaire. The school calendar of each participant will also be obtained.

Collection of Data

Sleep pattern will be monitored by actigraphy together with sleep diary throughout the whole study period. Twenty four-hour ambulatory BP monitoring and neurocognitive tests will be performed on the last day of each study week. All BP monitoring and neurocognitive tests will be performed during weekdays instead of weekends to avoid the possible weekend effect on sleep pattern and outcomes. Saliva samples will also be collected in the evening and the morning when the subjects are wearing the BP monitor for assessing cortisol awakening response.

Actigraphy

On day 1 of the first week of study, participants will attend our sleep laboratory to start actigraph recording (Actiwatch spectrum device; Phillips Respironics, Murrysville, PA; on their non-dominant wrist) and will be instructed on how to complete the sleep diary. Participants will have to wear the device until the end of the study period. Actigraphs will be configured to collect information in 1-minute epochs by using a medium sensitivity threshold, which has high sensitivity for detecting sleep compared with polysomnography. Self-reported bedtimes and wake times will be used to score actigraph data using established procedures. Variables of interest include actigraph-defined sleep period (ie, the period between scored sleep onset and scored final awakening), actigraph scored sleep (minutes of scored sleep within the actigraph-defined sleep period), wake after sleep onset (minutes of scored wake within the actigraph-defined sleep period), and sleep efficiency (actigraph scored sleep/actigraph-defined sleep period). The activity level during wakefulness will also be extracted as a covariate for statistical analysis, as it may affect both sleep pattern and BP.

Twenty four-hour ambulatory blood pressure monitoring

A validated oscillometric monitor (SpaceLabs 90217, SpaceLabs Medical, Redmond, Washington, USA) will be used. Systolic, diastolic and mean arterial BP will be measured every 30 minutes. The exact cut-off time dividing wake and sleep BP will be defined individually according to actigraphy. Recordings are included in the analysis when there is a minimum of 40 successful readings for the 24-hour period with a minimum of 1 successful reading per hour. Individual mean systolic, diastolic and mean arterial BP are calculated for wake and sleep periods. These BP data will be converted to z scores using the local "LMS" reference values (with reference to gender and height). Subjects will be defined as hypertensive if their systolic or diastolic BP is ≥95th percentile (z score ≥1.645).

Neurocognitive tests

Conners' Continuous Performance Test (CPT)

CPT-II (Ver. 5.2 for Windows®) is designed as a computer game-like test for the evaluation of sustained attention and response inhibition for respondents aged 6 or above. Subjects are required to press the space bar or click the mouse whenever any letter except the letter 'X' appears on the computer screen. The test requires about 14 minutes to complete, and it will be administered in the morning in a quiet room.

Trail-making Test Part A & B (Executive function)

The Trail-making test is composed of two parts which assess test-takers in attention, visual scanning, speed of eye-hand coordination, information processing and set switching of executive functions. Part A required subjects to connect sequentially 25 encircled numbers which are randomly scattered over the test sheet. Similarly, for Part B, subjects are asked connect encircled numbers (1-13) and alphabets (A-L) alternately in ascending patterns, i.e. 1-A-2-B-C. Any mistakes made throughout the test are pointed out by examiner immediately. Thus, the scores of the tests are the time taken to complete the task.

Stroop Test-Victoria Version (Executive function)

This test captures cognitive flexibility and inhibition of executive functioning by three successive tasks with increasing demands. It consists of three sets of stimulus cards (1) colored dots, (2) common words printed in same colors as dots, and (3) color words printed in non-corresponding colors of ink. For the first task, subjects are asked to simply name the color of the dots in maximum speed as possible. For the second task, subjects are asked to identify the color of ink each word is printed in, not to identify the word itself. For the third task, subjects are asked to identify the color of ink each of the color words is printed in, not to read the color word presented. Number of errors and time to perform the task are recorded for each trial. The Chinese Victoria Version of the Stroop Test is translated and validated by Dr. Tatia Lee and Dr. Kai Wang from the Laboratory of Neuropsychology, the University of Hong Kong.

Raven's Standard Progressive Matrices Test (Nonverbal reasoning)

The Test is a nonverbal measure of general ability that uses nonverbal stimuli including visual patterns and shapes to asses reasoning by analogy. It contains five sets with 12 problems in each set. Each question is a puzzle with a missing part; subjects are asked to identify the most appropriate piece from six similar options. Children of age 5 years 6 months to 8 years 5 months can do a shortened version with only Set A, B, and C to allow better control of test administration. Each set starts with a problem and develops a theme that build on previous questions and become progressively more difficult. The test is administered in a paper and pen format. While it is an open-ended session, most people complete the test in less than 40 minutes.

Grooved Pegboard (Visual-motor coordination)

It is a manipulative dexterity test aim at assessing visual-motor coordination. It consists of 25 holes with randomly positioned slots. Subjects are asked to place pegs, which have a key along one side, into the holes from left to right. The task is performed once with dominant hands and once with non-dominant hands. Subjects are advised to complete the task as fast as possible. Subjects from 5 years old to 8 years 12 months will use a Kiddie version of the test in which only the first two rows (10 pegs) of the pegboard are needed to complete. Time taken, number of pegs placed on the pegboard, and number of dropped pegs are recorded to assess the score of fine-motor coordination.

Cortisol awakening response (CAR)

Saliva samples will be collected with Salivette tubes for assessing the level of cortisol and cortisone, as a reflection of stress which on its own can influence both sleep pattern and BP.

Participants will be asked to collect their saliva in the morning. Each subject will have to provide five saliva samples according to a fixed sampling protocol: (1) one hour before bedtime, (2) immediately after awakening, (3) 15 min after awakening, (4) 30 min after awakening, and (5) 45 min after awakening. Salivary cortisol and cortisone concentrations in these samples will be measured by a liquid chromatography tandem mass spectrometry method at the Biomedical Mass Spectrometry Unit, Department of Chemical Pathology, Prince of Wales Hospital. Between-batch precision performance of the method has coefficients of variation of <5%. The lower limits of quantitation are <0.5 nmol/l.

ELIGIBILITY:
General inclusion criteria:

* Adolescents aged between 10-18 years;
* Written informed consent and assent obtained from parents and adolescents.

Inclusion criteria specific for the sleep deprived group:

* Self-reported time in bed (period from bedtime to get-up time) during school days of <8 hours per day
* Self-perceived insufficient sleep during school days

Inclusion criteria specific for the normal sleep group:

* Self-reported time in bed during school days of >=8 hours per day
* Self-perceived sufficient sleep during school days

Exclusion criteria

* Obesity which is defined as a body mass index (BMI) ≥95th percentile (corresponding to a z score of 1.645) of the local reference.
* Subjects who are having sleep disorder for example insomnia and/or currently receiving treatment for sleep problems.
* Known medical or psychiatric conditions or use of current medication that may affect sleep and BP.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Subjects will be recruited from local primary and secondary schools. We will send invitation letters to Principals to ask them for their help with screening questionnaire distribution and assessment arrangements in their school. The screening questionnaire asks about children sleep pattern during school terms and holidays, sleep-related symptoms (e.g. snoring), and medical history to see whether they are eligible to participate. Eligible subjects will receive the study factsheet and written informed consent form. Subjects with parental consent will be enrolled in our study.
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Change in ambulatory systolic blood pressure during wakefulness across school holidays | From 1 week before holiday to 1 week after holidays, an average of 4 weeks.
  Change in average systolic blood pressure during wakefulness as measured by 24-hour ambulatory blood pressure monitoring

SECONDARY OUTCOMES:
Changes in other ambulatory BP parameters | From 1 week before holiday to 1 week after holidays, an average of 4 weeks.
  Changes in average diastolic blood pressure during wakefulness, systolic blood pressure during sleep and diastolic blood pressure during sleep
Change in sleep duration | From 1 week before holiday to 1 week after holidays, an average of 4 weeks.
  Change in sleep duration measured by actigraphy
Change in vigilance | From 1 week before holiday to 1 week after holidays, an average of 4 weeks.
  Changes in vigilance measured by Conners' Continuous Performance Test (CPT)
Change in impulsivity | From 1 week before holiday to 1 week after holidays, an average of 4 weeks.
  Change in impulsivity measured by Conners' Continuous Performance Test (CPT)
Change in trail-making test score | From 1 week before holiday to 1 week after holidays, an average of 4 weeks.
  Change in executive function measured by trail-making test
Change in Stroop test score | From 1 week before holiday to 1 week after holidays, an average of 4 weeks.
  Change in executive function measured by Stroop test (Victoria Version)
Change in non-verbal reasoning | From 1 week before holiday to 1 week after holidays, an average of 4 weeks.
  Change in non-verbal reasoning measured by Raven's Standard Progressive Matrices Test
Change in visual-motor coordination | From 1 week before holiday to 1 week after holidays, an average of 4 weeks.
  Change in visual-motor coordination tested by Grooved Pegboard

CONTACTS AND LOCATIONS:
Overall Officials: Albert M Li, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Paediatrics, The Chinese University of Hong Kong, Hong Kong, Hong Kong

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-12): https://cdn.clinicaltrials.gov/large-docs/10/NCT03895710/Prot_SAP_000.pdf